CLINICAL TRIAL: NCT00632814
Title: A Prospective Study to Evaluate the Effect of rFVIII-FS in Different Prophylactic Regimens on Bleeding Events Frequency and Development of Arthropathy in Previously Treated and Minimally Treated Hemophilia A Pediatric Population.
Brief Title: Russian Kogenate Pediatric Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12684; 2014-005253-39 (EudraCT Number)
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hemophilia A
Keywords: Kogenate,; Children,; Factor VIII,; Hemophilia A,; Prophylactic
MeSH Terms: conditions — Hemophilia A | interventions — recombinant FVIII, sugar formulated; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw (Experimental): rFVIII-FS (Octocog-alfa, antihemophilic factor [recombinant]) 70 IU/kg, dosing by injection once per week [qw] (weekly on Day 7 + 1 after previous injection) for 9 months. Dose escalation was permitted due to joint bleeding (escalation to 35 IU/kg twice a week or further escalation to 25 IU/kg three times a week)
  Interventions: Drug: rFVIII-FS (Kogenate FS, BAY14-2222) 70 IU/kg, dosing once per week
- rFVIII-FS (Kogenate FS, BAY14-2222), biw (30 IU/kg + 40 IU/kg) (Experimental): rFVIII-FS (Octocog-alfa, antihemophilic factor [recombinant]) 70 IU/kg, dosing by injection twice per week [biw] (30 IU/kg [day 1] + 40 IU/kg [day 4]) for 9 months. Dose escalation was permitted due to joint bleeding (escalation to 25 IU/kg three times a week)
  Interventions: Drug: rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg twice per week (30 IU/kg + 40 IU/kg)
- rFVIII-FS (Kogenate FS, BAY14-2222), tiw (3 x 25 IU/kg) (Experimental): rFVIII-FS (Octocog-alfa, antihemophilic factor [recombinant]) 75 IU/kg, dosing by injection three times per week [tiw] (3 x 25 IU/kg [day 1, 3, 5]) for 9 months. No escalation opportunity for participants in this group
  Interventions: Drug: rFVIII-FS (Kogenate FS, BAY14-2222) 75 IU/kg, dosing three times per week (3 x 25 IU/kg)

INTERVENTIONS:
Drug: rFVIII-FS (Kogenate FS, BAY14-2222) 70 IU/kg, dosing once per week — rFVIII-FS (Octocog-alfa, antihemophilic factor [recombinant]) 70 IU/kg, dosing by injection once per week (weekly on Day 7 + 1 after previous injection) for 9 months. Dose escalation was permitted due to joint bleeding (escalation to 35 IU/kg twice a week or further escalation to 25 IU/kg three times a week)
  Arms: rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw
Drug: rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg twice per week (30 IU/kg + 40 IU/kg) — rFVIII-FS (Octocog-alfa, antihemophilic factor [recombinant]) 70 IU/kg, dosing by injection twice per week (30 IU/kg [day 1] + 40 IU/kg [day 4]) for 9 months. Dose escalation was permitted due to joint bleeding (escalation to 25 IU/kg three times a week)
  Arms: rFVIII-FS (Kogenate FS, BAY14-2222), biw (30 IU/kg + 40 IU/kg)
Drug: rFVIII-FS (Kogenate FS, BAY14-2222) 75 IU/kg, dosing three times per week (3 x 25 IU/kg) — rFVIII-FS (Octocog-alfa, antihemophilic factor [recombinant]) 75 IU/kg, dosing by injection three times per week (3 x 25 IU/kg [day 1, 3, 5]) for 9 months. No escalation opportunity for patients in this group
  Arms: rFVIII-FS (Kogenate FS, BAY14-2222), tiw (3 x 25 IU/kg)

SUMMARY:
A prospective study to evaluate the effect of rFVIII-FS in different prophylactic regimens on bleeding events frequency and development of arthropathy in Previously Treated and Minimally treated Hemophilia A pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Severe hemophilia A or moderate hemophilia A
* 1-12 years of age
* Requiring treatment with FVIII

Exclusion Criteria:

* Current or prior inhibitor or familial antecedents of inhibitor
* Surgery required during the study (9 months)
* Positive for HIV

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Russia (4):
  - Kirov
  - Moscow
  - Saint Petersburg
  - Yekaterinburg

REFERENCES:
- [Result] V.V. Vdovin, T.A. Andreeva, T.A. Chernova, F.G. Perina, E.E.M. Shiller, P.V. Svirin, M. Maas Enriquez, and S. Rauchensteiner. Prophylaxis with Once, Twice or Three-Times Weekly Dosing of rFVIII-FS Prevents Joint Bleeds in a Previously Treated Pediatric Population with Moderate/Severe Hemophilia A. Journal of Coagulation Disorders 2011; 3:(1). October 2011
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period took from first patient first visit 28 Jun 2007 to last patient first visit 26 Dec 2008. The study period took from first patient first visit 28 Jun 2007 to last patient last visit 27 Sep 2009. All 4 sites were medical clinics. Assignment to a group was based on patients previous treatment schedule (non-randomized).
Pre-assignment Details: There was an indefinite time period between screening and baseline. Study treatment started at visit 2 (baseline).
Period: Overall Study
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Started | 11 | 13 | 8
Completed | 11 | 13 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg) | Total
Number analyzed (Participants) | 11 | 13 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.27 (3.20) | 6.08 (3.50) | 6.00 (3.12) | 5.09 (3.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 11 | 13 | 8 | 32
Ethnicity [Number; unit: participants]
  Caucasian | 11 | 13 | 7 | 31
  Asian | 0 | 0 | 1 | 1
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 17.48 (10.43) | 24.39 (11.35) | 25.45 (9.87) | 22.28 (10.93)
Height [Mean (Standard Deviation); unit: Centimeters] | 98.09 (22.88) | 120.31 (23.75) | 122.00 (20.74) | 113.09 (24.63)
Number of participants on Prophylaxis Prior to Screening [Number; unit: pariticipants] — Number of participants on prophylaxis versus on-demand therapy before screening
  pariticipants
    On demand | 9 | 6 | 5 | 20
    Prophylaxis | 2 | 7 | 3 | 12
FVIII trough level at Baseline [Mean (Standard Deviation); unit: Percentage of FVIII activity] | 1.43 (0.70) | 1.62 (1.79) | 0.77 (0.24) | 1.34 (1.24)
Number of participants with different exposure days (ED) [Number; unit: participants]
  0 ED | 1 | 0 | 0 | 1
  1 to <20 ED | 1 | 0 | 0 | 1
  20 to <100 ED | 4 | 2 | 4 | 10
  >=100 ED | 5 | 11 | 4 | 20
Percentage of participants with Target Joint Present [Number; unit: Percentage of participants] | 36 | 54 | 88 | 178
Number of participants with bleeding rates in previous 6-9 Months [Number; unit: participants]
  No bleedings | 1 | 2 | 0 | 3
  Any bleedings | 10 | 11 | 8 | 29
  Any joint bleedings | 9 | 11 | 6 | 26
Stockholm Joint Score [Mean (Standard Deviation); unit: scores on a scale] — The assessment of joint function using Stockholm Joint Score. The minimum value is 0 (the best condition), and the maximum value is 140 (the worst condition).
  scores on a scale | 3.9 (4.8) | 5.9 (5.8) | 7.1 (4.6) | 5.5 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Less Than 2 Joint Bleeds During the 9-month Treatment Period
Time Frame: Up to 9 months
Measure: Number; unit: Percentage of participants
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
Percentage of participants | 72.7 | 84.6 | 75.0

2. Secondary Outcome: Number of Bleeds Per Participant During the 9-month Treatment Period
Time Frame: Up to 9 months
Measure: Median (Full Range); unit: bleeds per participant
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
bleeds per participant
  All bleeds | 3.0 [0 to 12] | 2.0 [0 to 6] | 1.5 [0 to 8]
  Joint bleeds | 0 [0 to 2] | 0 [0 to 3] | 0 [0 to 8]

3. Secondary Outcome: Number of Participants With Bleeding Events During the 9-month Treatment Period
Time Frame: Up to 9 months
Measure: Number; unit: Participants
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
Participants
  no bleeds | 3 | 4 | 4
  bleeds at all | 8 | 9 | 4

4. Secondary Outcome: Number of Participants With Joint Bleeds During the 9-month Treatment Period
Time Frame: Up to 9 months
Measure: Number; unit: Participants
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
Participants
  no bleeds | 8 | 9 | 6
  bleeds at all | 3 | 4 | 2

5. Secondary Outcome: Number of Participants in Each Group at the End of the Study
Time Frame: Up to 9 months
Population: Participants were allowed to switch treatment groups upon occurrence of joint bleed. Therefore the number of participants per group at the end of the study is different from the number of participants per group at baseline.
Measure: Number; unit: Participants
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
Participants | 8 | 14 | 10

6. Secondary Outcome: Actual Monthly rFVIII-FS Consumption
Time Frame: Up to 9 months
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
IU/kg | 390.8 (106.9) | 422.3 (138.2) | 501.4 (241.2)

7. Secondary Outcome: Change From Baseline in Stockholm Hemophilia Joint Score at 9 Months of Treatment
Description: The assessment of joint function using Stockholm Joint Score. The minimum value is 0 (the best condition), and the maximum value is 140 (the worst condition).
Time Frame: baseline and 9 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 11 | 13 | 8
Scores on a scale | -1.4 (2.4) | -2.0 (4.5) | -1.8 (2.2)

8. Secondary Outcome: Haemo-QoL Standardized Total Score at 9 Months of Treatment (Completed by Participants in the Total Group)
Description: Quality of life (QoL) was measured by the Haemo-QoL standardized total Score, which ranged from 0 (the best condition) to 100 (the worst condition).
Time Frame: 9 months
Population: Participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 3 | 10 | 7
Scores on a scale | 30.28 (13.09) | 39.07 (23.50) | 30.27 (11.95)

9. Secondary Outcome: Haemo-QoL Standardized Total Score (Completed by Parents/Caregivers in the Total Group) at 9 Months of Treatment
Description: as for outcome 8
Time Frame: 9 months
Population: Participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Number analyzed (Participants) | 3 | 10 | 7
Scores on a scale | 29.13 (17.40) | 28.43 (10.27) | 31.38 (13.06)

ADVERSE EVENTS:
Arm/Group | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg)
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/13 | 0/8
Other Adverse Events (participants affected / at risk) | 4/11 | 3/13 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw (N=11) | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) (N=13) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg) (N=8)
Factor VIII inhibition (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFVIII-FS (Kogenate FS, BAY14-2222), 70 IU/kg qw (N=11) | rFVIII-FS (Kogenate FS, BAY14-2222), Biw (30 IU/kg + 40 IU/kg) (N=13) | rFVIII-FS (Kogenate FS, BAY14-2222), Tiw (3 x 25 IU/kg) (N=8)
Adenoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Yersinia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (4)

LIMITATIONS AND CAVEATS:
Protocol deviations were not excluded: e.g. a previously untreated patient developed the transitory inhibitor; change to a higher group did not always occur according protocol; there was temporary lack of smaller vial sizes at the centers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institute shall supply a draft of any intended publication to the Customer not less than 60 (sixty) days before submission it for the publication in question and will supply a draft of any abstract or detailed paper or oral statement intended for public presentation not less than 60 (sixty) days before the earliest of the date of submission of the abstract or delivery of the public presentation. The Institute agrees that in any such publication only such data as is contained in an analysis.